CLINICAL TRIAL: NCT03454659
Title: Comparison of the Effect of Low and High Fraction of Inspired Oxygen on Postoperative Surgical Field Infection and Pulmonary Complications in Patients Undergoing Supratentorial Craniotomy
Brief Title: Comparison of the Effect of Low and High Fraction of Inspired Oxygen on Postoperative Surgical Field Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Aydın, Research Assistant, Istanbul University
Other Study IDs: 83045809-604.01.02-
Record Dates: First submitted 2018-01-17; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Supratentorial Brain Tumor
MeSH Terms: interventions — Craniotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high (0.8 ): The purpose of this study is to compare the effect of high 0.8 and low 0.4 FiO2 ventilation primarily on surgical field infection and secondarily on postoperative pulmonary complications in patients are undergoing supratentorial craniotomy surgeons.
  Interventions: Procedure: Craniotomy
- low (0,4) fiO2: The purpose of this study is to compare the effect of high 0.8 and low 0.4 FiO2 ventilation primarily on surgical field infection and secondarily on postoperative pulmonary complications in patients undergoing supratentorial craniotomy surgeons.
  Interventions: Procedure: Craniotomy

INTERVENTIONS:
Procedure: Craniotomy — Extracting the part of the sculpt

SUMMARY:
The purpose of this study is to compare the effect of high 0.8 and low 0.4 *FiO2 ventilation primarily on surgical field infection and secondarily on postoperative pulmonary complications in patients are undergoing supratentorial craniotomy surgeons.

*fraction of inspired oxygen

DETAILED DESCRIPTION:
The aim of the study is to compare effects of high 0.8 FiO2 and low 0.4 FiO2 in patients are undergoing supratentorial craniotomy surgery primarily on postoperative surgical wound infection and secondarily on postoperative pulmonary complications.

The study will be performed prospectively in patient are undergoing elective supratentorial craniotomy with supine position at Istanbul university Cerrahpasa Medical School Department of Neurosurgery operating room. ASA class I-III 80 patients will be included the study. Exclusion criteria are obstructive or restrictive lung disease, chest wall deformity, congestive heart failure, liver or kidney failure, postoperatively non-cooperative and unconsciousness, preoperative fever and infection history, serious malnutrition( plasma albumin level < 3 g/dl, WBC <2500/mm3 or weight loss more than 20% in 3 months),and diabetes mellitus.

The gender, age, height, weight, BMI, smoking history and systemically illness of patients will be recorded. Patients will be randomized with closed envelop technique and divided in 2 groups. All patients will be monitored ECG, heart rate, invasive blood pressure , FiO2,pulse oximetry (SpO2) and end tidal carbon dioxide . Propofol (2 mg kg-1), remifentanyl (0.15 µ kg-1), rocuronium (0.6 mg kg-1) will be used for induction in both groups. Anesthesia maintenance will be provided with sevoflurane (1 MAC), remifentanyl (0.05-0.1 µ kg-1 dk-1) and rocuronium (0.3 mg kg-1 sa-1) . Patients will be intubated orotracheally and ventilated with volume control mode ( tidal volume 8 mL/kg, respiratory frequency will be adjusted between 9-12/minutes to hold PaCO2 between 33-35 mmHg ,inspiration/expiration ratio ½,PEEP:5 cmH2O ). Peroperative analgesia will be provided with remifentanyl infusion. Ondansetron 8 mg for antiemesis and tramadol 100 mg for postoperative analgesia will be administered intravenously 30 minutes before extubation. Duration of surgery and non-invasive cerebral oxygen saturation (SctO2) using bilateral frontal electrodes will be recorded. At the end of the surgery, sugammadex 2mg kg-1 will be administered for decurarization in all groups. Patients will be transferred to the recovery room in postoperative period and 15L/min and 4L/min oxygen will be given to 0.8 FiO2 group and other group, respectively.

Wound healing will be evaluated every day in terms of surgical wound infection occurrence for postoperative 14 days with ASEPSIS classification. Surgical wound infection will be considered in patients who score 20 or more on daily basis. The patients who are discharged will be reached by phone. Pneumonia, atelectasis, respiratory failure, hospital and intensive care unit stay will be recorded for postoperative 14 days. *CDC criteria will be used to diagnose pneumonia. Respiratory insufficiency is diagnosed by SpO2 fall below 90% despite oxygen treatment and mechanical ventilation need. If pulmonary complication develops ,findings will be recorded with chest radiography or tomography when necessary.

* ASA: american society of anaesthesiology
* WBC:white blood cell
* PEEP: positive end expiratory pressure
* CDC: centers for disease control and prevention

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-3

Exclusion Criteria:

* Obstructive and restrictive lung disease
* Chest wall deformity
* Chronical heart failure
* Liver and kidney failure
* Preoperative fever and infection history
* Important malnutrition
* Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * ASA CLASS 1-3
  * Patient age between 18-70 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
the rate of surgical field infection will be evaluated by ASEPSIS score. | 2 years
  Table 1 ASEPSIS SCORE. Proportion of wound affected (%) Wound characteristic 0 <20 20-39 40-50 60-79 >80
  Serous exudate 0 1 2 3 4 5 Erythema 0 1 2 3 4 5 Purulent exudate 0 2 4 6 8 10 Separation of deep tissues 0 2 4 6 8 10
  Criterion Points Additional treatment Antibiotics 10 Drainage of pus under local anesthesia 5 Debridement of wound (general anaesthesia) 10 Serous discharge daily 0-5 Erythema daily 0-5 Purulent exudate daily 0-10 Separation of deep tissues daily 0-10 Isolation of bacteria 10 Stay as inpatient prolonged over 14 days 5
  Total score Infection category 0-10 Satisfactory healing 11-20 Disturbance of healing 21-30 Minor wound healing 31-40 Moderate wound infection. >40 Severe wound infection

SECONDARY OUTCOMES:
The rate of postoperatively pulmonary complications such as pneumonia,respiratory failure will be evaluated.Centers for Disease Control and Prevention criteria will be used for defining nosocomial pneumonia. | 2 years
  The diagnosis of respiratory failure will be perform by reduction of SpO2 ≤ 90% although oxygen treatment and/or need for noninvasive or invasive mechanical ventilation.

REFERENCES:
- See also: High-concentration supplemental perioperative oxygen to reduce the incidence of postcesarean surgical site infection: a randomized controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/18757651
- See also: New WHO recommendations on intraoperative and postoperative measures for surgical site infection prevention: an evidence-based global perspective. — http://www.ncbi.nlm.nih.gov/pubmed/27816414
- See also: Wound hypoxia and acidosis limit neutrophil bacterial killing mechanisms. — http://www.ncbi.nlm.nih.gov/pubmed/9301612
- See also: WHO Needs High FIO2? — http://www.ncbi.nlm.nih.gov/pubmed/28868164
- See also: Oxygen concentration and characteristics of progressive atelectasis formation during anaesthesia. — http://www.ncbi.nlm.nih.gov/pubmed/21039356
- See also: Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. — http://www.ncbi.nlm.nih.gov/pubmed/19826023